CLINICAL TRIAL: NCT05242939
Title: Comparison of Active and Passive Distraction Techniques in Reducing Anxiety and Fear Levels During Inhalation Therapy in Children: A Randomized Controlled Study
Brief Title: Active and Passive Distraction Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Uğur Gül, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Inhalation Therapy in Children
Record Dates: First submitted 2021-12-28; First posted 2022-02-16 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Child, Only; Inhalation Therapy; Complications
Keywords: inhalation therapy; child; fear; cartoon; video game

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Group of Cartoons (Experimental): The cartoons that are suitable for the child's age and gender will be watched. The child will be asked which cartoon he would like to watch. The cartoon is 5 min from the application. It will be started to be watched first and will continue until the application is finished. Vital signs (pulse, respiration and SPo2), Child Fear Scale and Child Anxiety Scale-State Statement Scale (CAS-D) will be evaluated by the researcher and the child before, immediately and 5 minutes after the application and recorded in the intervention follow-up form by the researcher. Due to the COVID-19 pandemic, cartoons will be watched on the parent's phone. Parents who do not have an internet connection will also be provided with internet access by the researcher. The child will watch cartoons on their parent's phone.
  Interventions: Other: Watching cartoons
- The Group of Game (Experimental): 723 / 5.000 Çeviri sonuçları The group whose video games will be played will be told to choose the game they want before the process. Due to the COVID-19 pandemic, video games will be played on the parent's phone. Parents who do not have an internet connection will also be provided with internet access by the researcher. The child will play the video game on their parent's phone.
  Interventions: Other: Video game
- Rutin Care Group (No Intervention): In the control group, the institution's routine nebula application will be performed and no intervention will be made. Vital signs (pulse, respiration and SPo2), Child Fear Scale and Child Anxiety Scale-State Statement Scale (CAS-D) will be evaluated by the researcher and the child before, immediately and 5 minutes after the application and recorded in the intervention follow-up form by the researcher.

INTERVENTIONS:
Other: Video game — The child will be allowed to play the game they want to play throughout the entire procedure, starting 5 minutes before the inhalation therapy. Vital signs (pulse, respiration and SPo2), Child Fear Scale and Child Anxiety Scale-State Statement Scale (CAS-D) will be evaluated by the researcher and the child before, immediately and 5 minutes after the application and recorded in the intervention follow-up form by the researcher.
  Arms: The Group of Game
Other: Watching cartoons — The cartoon is 5 min from the application. It will be started to be watched first and will continue until the application is finished. Vital signs (pulse, respiration and SPo2), Child Fear Scale and Child Anxiety Scale-State Statement Scale (CAS-D) will be evaluated by the researcher and the child before, immediately and 5 minutes after the application and recorded in the intervention follow-up form by the researcher.
  Arms: The Group of Cartoons

SUMMARY:
Treatment methods with nebulizers are used in the treatment of many diseases such as asthma, bronchitis, bronchiolitis and cystic fibrosis in children. Because inhalation therapy with a face mask is scary for children, it can be difficult to provide this therapy effectively and safely. Adaptation of the child and family is important for the success of inhalation therapy. Distraction techniques are among the most commonly used cognitive/behavioral methods. It determines the effect of "playing video games" and "watching cartoons" methods, which are active distraction methods during inhalation therapy, on the level of fear and anxiety.

DETAILED DESCRIPTION:
Hospitalization can be a threatening and stressful experience for children. Unfamiliar with the environment and medical procedures and unaware of the reasons for hospitalization can result in children's anger, uncertainty, anxiety and feelings of helplessness. Anxiety and fear are the most frequently reported among these negative reactions. In addition, high levels of anxiety and fear can be harmful to children's physiological and psychological health. Excessive anxiety and fear also inhibit children's effectiveness in coping with medical treatment and increase their negative emotions. It is thought that the levels of anxiety and fear in children will increase even more when they apply to the emergency services, especially in acute situations. Children who present to the emergency department with respiratory distress and cough can be given inhalation therapy as a result of physical examination and other tests. Today, inhalation therapy with a nebulizer is one of the most common and frequently used methods. Treatment methods with nebulizers are used in the treatment of many diseases such as asthma, bronchitis, bronchiolitis and cystic fibrosis in children. Because inhalation therapy with a face mask is scary for children, it can be difficult to provide this therapy effectively and safely. Adaptation of the child and family is important for the success of inhalation therapy.

Evidence-based distraction methods can be used to provide effective inhalation and reduce fear of children. Recent research has focused on the use of non-pharmacological methods in the management of pain in children. Non-pharmacological methods used to manage pain and anxiety in children fall into three main groups; supportive methods, cognitive/behavioral methods, and physical methods. Distraction techniques are among the most commonly used cognitive/behavioral methods. It has been reported that distraction cards, watching cartoons, using kaleidoscope, and listening to music reduce pain, anxiety and fear levels. It is noteworthy that similar studies mostly focused on invasive applications. On the other hand, it is stated that studies on the effect of non-pharmacological methods in inhalation therapy, which is one of the common non-invasive procedures in children, are still limited. Another aim of this study is; This study determines the effect of "playing video games" and "watching cartoons" methods, which are active distraction methods during inhalation therapy, on the level of fear and anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 4-7 years
2. Children who have not undergone any painful procedures before the procedure
3. Parents with smartphones
4. Children and parents who can speak and understand Turkish
5. Children of parents who agreed to participate in the study and whose written consent form was obtained from them will be included in the study.

Exclusion Criteria:

1. Having a neurological disorder,
2. Congenital anomaly,
3. Growth and development retardation,
4. Hearing impaired,
5. Having visual impairment,
6. Having a chronic disease,
7. Using anti-epileptic drugs in the last 6 hours,
8. Children with suspected COVID-19 will not be included in the study.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-02-19 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Child Fear Scale (CFS) Measure | 1 year
  The Child Fear Scale is aimed at children between the ages of 4-10 and was used to evaluate the anxiety in children before and during the procedure. The CLS, which was translated into Turkish by Gerceker et al. (2018) and whose validity and reliability studies were conducted in Turkish, was developed by McKinley et al. The mean score of the CLS, which was translated into Turkish by five independent linguists, was 1.9 ± 0.1 (min=0, max=4). CLS can also be scored by parents and researchers. The CLS consists of five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety).
  The Child Fear Scale score will be recorded five minutes before the intervention, during intervention and five minutes after intervention
Child Anxiety Scale-State (CAS-S) | 1 year
  The Child Anxiety Scale-Status (CAS-S) scale, developed by Ersig et al. to measure the anxiety levels of children aged 4-10. Validity and reliability study was conducted for children aged 10 years, and the validity index was found to be 1.00 for the Child Anxiety Scale-State Scale.The ÇAS-S scale is similar to a thermometer with a light bulb at the bottom and horizontal lines at intervals that go up. On this scale for 4-10 year olds, children may say, "Imagine all your anxious or angry feelings are on the bulb or the bottom of the thermometer" or "If you're a little worried or nervous, emotions may run a little higher on the thermometer. If you are very, very anxious or nervous, the emotions can run high. Put a line on the thermometer to show how worried or angry you are." In order to measure state anxiety (CAS-S), the child is asked to mark what he feels "at the moment". The score can vary between 0 - 10.

SECONDARY OUTCOMES:
Pulse oximetry | 1 year
  Pulse oximetry is a portable monitor that displays peak heart rate and oxygen saturation values together. Heartbeat will be checked with the Nellcor device attached to the baby's right index finger. Pulse oximetry score will be recorded five minutes before the intervention, during intervention and five minutes after intervention
Heartbeat | 1 year
  Heartbeat will be checked with the Nellcor device attached to the baby's right index finger.
  Heratbeat score will be recorded five minutes before the intervention, during intervention and five minutes after intervention
Respiratory | 1 year
  Participant's respiration will be measured by the researcher. Respiratory score will be recorded five minutes before the intervention, during intervention and five minutes after intervention
Spo2 | 1 year
  Spo2 will be checked with the Nellcor device attached to the baby's right index. Spo2 score will be recorded five minutes before the intervention, during intervention and five minutes after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Uğur Gül, Principal Investigator — Akdeniz Univercity
Locations (1):
- Akdeniz University, Kepez, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alhaider SA, Alshehri HA, Al-Eid K. Replacing nebulizers by MDI-spacers for bronchodilator and inhaled corticosteroid administration: Impact on the utilization of hospital resources. Int J Pediatr Adolesc Med. 2014 Sep;1(1):26-30. doi: 10.1016/j.ijpam.2014.09.002. Epub 2014 Oct 22. PMID 32289071
- [Background] Amirav I, Newhouse MT, Minocchieri S, Castro-Rodriguez JA, Schuepp KG. Factors that affect the efficacy of inhaled corticosteroids for infants and young children. J Allergy Clin Immunol. 2010 Jun;125(6):1206-11. doi: 10.1016/j.jaci.2010.01.034. Epub 2010 Mar 24. PMID 20338620
- [Background] Ari A, Fink JB. Guidelines for aerosol devices in infants, children and adults: which to choose, why and how to achieve effective aerosol therapy. Expert Rev Respir Med. 2011 Aug;5(4):561-72. doi: 10.1586/ers.11.49. PMID 21859275
- [Background] Aydin D, Sahiner NC, Ciftci EK. Comparison of the effectiveness of three different methods in decreasing pain during venipuncture in children: ball squeezing, balloon inflating and distraction cards. J Clin Nurs. 2016 Aug;25(15-16):2328-35. doi: 10.1111/jocn.13321. Epub 2016 Apr 26. PMID 27112434
- [Background] Fernandes SC, Arriaga P. The effects of clown intervention on worries and emotional responses in children undergoing surgery. J Health Psychol. 2010 Apr;15(3):405-15. doi: 10.1177/1359105309350231. PMID 20348361
- [Background] DiBlasi RM. Clinical Controversies in Aerosol Therapy for Infants and Children. Respir Care. 2015 Jun;60(6):894-914; discussion 914-6. doi: 10.4187/respcare.04137. PMID 26070582
- [Background] Durak H, Uysal G. The Effect of Cartoon Watching and Distraction Card on Physiologic Parameters and Fear Levels During Inhalation Therapy in Children: A Randomized Controlled Study. J Trop Pediatr. 2021 Jan 29;67(1):fmab018. doi: 10.1093/tropej/fmab018. PMID 33742204
- [Background] Ersig AL, Kleiber C, McCarthy AM, Hanrahan K. Validation of a clinically useful measure of children's state anxiety before medical procedures. J Spec Pediatr Nurs. 2013 Oct;18(4):311-9. doi: 10.1111/jspn.12042. Epub 2013 Jun 25. PMID 24094126
- [Background] Tufekci FG, Celebioglu A, Kucukoglu S. Turkish children loved distraction: using kaleidoscope to reduce perceived pain during venipuncture. J Clin Nurs. 2009 Aug;18(15):2180-6. doi: 10.1111/j.1365-2702.2008.02775.x. PMID 19583650
- [Background] Kwok PC, Chan HK. Delivery of inhalation drugs to children for asthma and other respiratory diseases. Adv Drug Deliv Rev. 2014 Jun;73:83-8. doi: 10.1016/j.addr.2013.11.007. Epub 2013 Nov 21. PMID 24270011
- [Background] Mutlu B, Balci S. Effects of balloon inflation and cough trick methods on easing pain in children during the drawing of venous blood samples: a randomized controlled trial. J Spec Pediatr Nurs. 2015 Jul;20(3):178-86. doi: 10.1111/jspn.12112. Epub 2015 Mar 28. PMID 25817062
- [Background] Risaw L, Narang K, Thakur JS, Ghai S, Kaur S, Bharti B. Efficacy of Flippits to Reduce Pain in Children during Venipuncture - A Randomized Controlled Trial. Indian J Pediatr. 2017 Aug;84(8):597-600. doi: 10.1007/s12098-017-2335-z. Epub 2017 Apr 5. PMID 28378139
- [Result] Inan G, Inal S. The Impact of 3 Different Distraction Techniques on the Pain and Anxiety Levels of Children During Venipuncture: A Clinical Trial. Clin J Pain. 2019 Feb;35(2):140-147. doi: 10.1097/AJP.0000000000000666. PMID 30362982
- See also: Effectiveness Of '' Animated Cartoons '' As A Distraction Strategy On Behavior Response To Pain Perception Among Children Undergoing. Venipuncture — https://nrfninechd.com/effectiveness-of-animated-cartoons-as-a-distraction-strategy-on-behavior-response-to-pain-perception-among-children-undergoing-venipuncture/
- See also: The Effect of Distraction Technique on the Pain of Dressing Change among 3-6 Year-old Children — https://ijp.mums.ac.ir/article_6699_54b321fedd9302a43ce53253b6115a47.pdf
- See also: Durumluk-sürekli kaygı envanteri el kitabı — https://www.worldcat.org/title/durumluk-surekli-kayg-envanteri-el-kitab/oclc/81840585
- See also: Effects of Distraction on Physiologic Indices and Pain Intensity in children aged 3-6 Undergoing IV Injection — https://eds.p.ebscohost.com/eds/pdfviewer/pdfviewer?vid=0&sid=66b76973-d10b-4e04-9fd8-5b00941ee69a%40redis
- See also: Primary out come — https://dergipark.org.tr/tr/download/article-file/752838